CLINICAL TRIAL: NCT03683069
Title: Hypertension and Striatin Gene Structure Related to Aldo Phenotype
Brief Title: Mineralocorticoid Receptor (MR) Antagonist (Eplerenone) vs Amlodipine and STRIATIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Gordon H. Williams, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2018P001888; R01HL144779 (NIH)
Record Dates: First submitted 2018-09-17; First posted 2018-09-25 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Genetics Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Parallel Design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The screened, eligible hypertensives will enter a two-week single blind placebo washout phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eplerenone Arm (Experimental): antihypertensive eplerenone
  Interventions: Drug: Eplerenone vs Amlodipine
- Amlodipine Arm (Experimental): antihypertensive amlodipine
  Interventions: Drug: Eplerenone vs Amlodipine

INTERVENTIONS:
Drug: Eplerenone vs Amlodipine — We posit that decreases in striatin activity/levels increases aldosterone secretion resulting in hypertension and salt sensitive blood pressure. Thus, our mechanistic clinical study will assess whether hypertensive striatin risk allele carriers will show significantly greater reductions in blood pressure with a specific aldosterone mediated treatment approach (mineralocorticoid receptor blockade) than with a non-specific approach (amlodipine). To test this hypothesis, we will perform a randomized, double-blind, active controlled study in hypertensive carriers of the striatin risk allele using a novel two-limb, proof-of-principle study. Our primary outcome will be a liberal salt diet systolic blood pressure with a secondary outcome of salt sensitive blood pressure. Therefore, this mechanistic trial will provide support for using a genetic marker that identifies individuals who are uniquely responsive to mineralocorticoid receptor blockade--personalized, precision medicine.

SUMMARY:
Salt sensitivity of blood pressure is a substantial risk factor for cardiovascular morbidity and mortality. Inappropriate increases in renal sodium reabsorption lead to volume expansion, hypertension and salt sensitive blood pressure. Key homeostatic mechanisms that regulate renal sodium reabsorption are: first, hormonal, e.g., renin-angiotensin-aldosterone system and second, vascular, e.g., renal vasculature. Dysfunction in one or both mechanisms leads to hypertension and salt sensitive blood pressure. The investigators recently documented that striatin plays a novel role in the development of salt sensitive blood pressure. However, the mechanisms that lead to striatin-mediated salt sensitive blood pressure are not clear; defining these mechanisms is the overall goal of this proposal.

Striatin is a calmodulin- and caveolin-binding protein that can function as either a scaffolding and/or signaling protein, specifically in relation to the mechanism of action of steroids. In a large study of well characterized subjects from the International Hypertensive Pathotype (HyperPATH) cohort, the investigators documented that hypertensive and normotensive humans who are striatin risk allele carriers have salt sensitive blood pressure.

The investigators then developed a striatin heterozygous knockout mouse as a tool to identify potential mechanisms for the salt sensitive blood pressure. The investigators documented that these mice also have salt sensitive blood pressure with higher blood pressure levels and inappropriately increased aldosterone levels on a liberal salt diet.

DETAILED DESCRIPTION:
HYPOTHESIS:

Hypertensive striatin risk allele carriers will show significantly greater reductions in blood pressure with a specific aldosterone mediated treatment approach (mineralocorticoid receptor blockade) than with a non-specific approach (amlodipine).

PROTOCOL:

1. The screened, eligible hypertensives will enter a two to three-week single blind placebo washout phase. Pill count will be used to determine compliance. Those with blood pressure between 145-170/90-109 mmHg and pill count between 80-100% after two to three-weeks will enter the randomized phase and counseled regarding salt intake.
2. The first step: subjects will be fed a 10 mEq Na+, 100 mEq K+ calculated diet for 6 days. The meals will be provided by the CCI Dietary Core. On the 7th day, the subjects will come to the CCI Ambulatory Clinical Center. After remaining supine for 60-90 minutes, the subjects will have blood samples obtained for future analyses and their blood pressure measured using an automatic recording sphygmomanometer (Space Labs, Snoqualmie, WA). Readings will be obtained every 2 minutes for 20 minutes with the highest and lowest values discarded and the rest averaged. From the morning of the 6th to the morning of the 7th day, a 24-hr. urine will be collected for creatinine and sodium as a check on balance and stored for future analyses.
3. The second step: Subjects will be counseled regarding liberal salt dietary intake. Subjects will be given high salt broth packets, calcium tablets (as calcium bicarbonate), and potassium tablets (as potassium bicarbonate) to supplement their diet to ensure similar intakes in all subjects [Na+ (200 mEq), potassium (K+, 100 mEq) and calcium (800 mg)]. This or a greater level of Na+ intake was consumed by 60-70% of subjects before entering the HyperPATH protocol. On the morning of the 6th day the subject will begin a 24-hour blood pressure recording, using a blood pressure machine provided by study staff. After completion of this diet for 6 days, the subject will come to the Center for Clinical Investigation (CCI) Ambulatory Clinical Center and after remaining supine for 60-90 mins will have blood samples obtained for future analyses, and their BP measured using an automatic recording sphygmomanometer (Space Labs, Snoqualmie, WA). Readings will be obtained every 2 mins for 20 mins with the highest and lowest values discarded and the rest averaged. From the morning of the 6th to the morning of the 7th day, a 24-hr. urine will be collected for creatinine and Na+ as a check on balance and stored for future analyses. The BP data from 2) and 3) will allow us to calculate Salt Sensitivity of Blood Pressure (SSBP), an approach performed successfully more than 500 times in the HyperPATH cohort.
4. The hypertensive striatin risk carrier subjects will be randomized, double blinded to one of two primary treatment groups and titrated to effect every four weeks, as was previously reported (1, 2), eplerenone 50, 100 and 200 mg daily or amlodipine 2.5, 5 and 10 mg daily. Study duration will be sixteen weeks.
5. Participants will be randomized in blocks of four to 1 of 2 study drugs (amlodipine and eplerenone). The drug class assignment will remain the same throughout the study for each subject. The PI or Co-PI will notify The Brigham and Womens Hospital Investigational Drug Pharmacy Service to escalate or maintain current dose on each of the two visits. The Brigham and Womens Hospital Investigational Drug Pharmacy Service will be responsible for the randomization schema, recording of study drug assignment, and dispensing of prescriptions. All others (PI, Co-PI, research staff, subject) will be blinded as to drug assignment.
6. Home seated, morning cuff blood pressure and pulse will be obtained daily and monitored by study staff weekly as a safety check with the information provided to the study staff by email or phone. The blood pressure results from the 7 days prior to the next visit will be averaged, with the highest and lowest values discarded. This average blood pressure value will be used to determine if the drug dose will be titrated after the next visit If the subject has reached goal blood pressure (less than or equal to140/90 mmHg), then the subject is maintained on his/her current dose. If not, the subject's dose is up titrated as per protocol. A member of the research team will contact the subject if the blood pressure data are not received within 24-hr of the designated time. If the cuff blood pressure is greater than 170/109 mmHg on two consecutive occasions 24 hours apart, or the subject develops cardiovascular symptoms, the subject will be terminated from the study and re-started on medications used before the washout period. The subject's physician will be contacted.
7. Because eplerenone may increase Serum K+ levels, we will monitor its level monthly during the study. This will be obtained at the time of their monthly visit unless a dose increase is made at the time of the visit. Then, the Serum K+ will be obtain one week later. If Serum K+ is greater than 5.5 milliMolar (mM) on two consecutive occasions 24 hours apart, the subject will be terminated from the study. If unexpected adverse event is noted The Brigham and Women's Hospital Investigational Drug Pharmacy Service will be notified so as to break code and identify agent.
8. At the end of four weeks since randomization and the subjects have completed the first dose of the agent, the subject will be counseled regarding a 24-hour dietary intake of sodium (200 mEq), potassium (100 mEq) and calcium (800 mg). Subjects will receive supplementary high salt broth packets to ensure that they are reaching the target Na+ intake. After completion of this diet for 6 days, the subject returns to Center for Clinical Investigation - Ambulatory Clinical Center and after remaining supine for 60-90 minutes again will have blood samples obtained for future analyses and their blood pressure measured using an automatic recording sphygmomanometer. Readings will be obtained every 2 minutes for 20 minutes with the highest and lowest values discarded and the rest averaged. This measurement will be used to assess the blood pressure response to a single dose of each agent. From the morning of the 6th to the morning of the 7th day, a 24-hr. urine will be collected for creatinine and sodium as a check on balance and stored for future analyses.
9. Home seated, morning cuff blood pressure and pulse will be obtained daily and monitored by study staff weekly as a safety check with the information provided to the study staff by email or phone. The blood pressure results from the 7 days prior to the next visit will be averaged, with the highest and lowest values discarded. This average blood pressure value will be used to determine if the drug dose will be titrated after the next visit If the subject has reached goal blood pressure (less than or equal to140/90 mmHg), then the subject is maintained on his/her current dose. If not, the subject's dose is up titrated as per protocol. A member of the research team will contact the subject if the blood pressure data are not received within 24-hr of the designated time. If the cuff blood pressure is greater than 170/109 mmHg on two consecutive occasions 24 hours apart, or the subject develops cardiovascular symptoms, the subject will be terminated from the study and re-started on medications used before the washout period. The subject's physician will be contacted.
10. Because eplerenone may increase Serum K+ levels, we will monitor its level monthly during the study. This will be obtained at the time of their monthly visit unless a dose increase is made at the time of the visit. Then, the Serum K+ will be obtain one week later. If Serum K+ is greater than 5.5 mM on two consecutive occasions 24 hours apart, the subject will be terminated from the study. If unexpected adverse event is noted The Brigham and Women's Hospital Investigational Drug Pharmacy Service will be notified so as to break code and identify agent.
11. At the end of eight weeks since randomization and the subjects have completed the second dose of the agent, the subject will be counseled regarding a 24-hour dietary intake of sodium (200 mEq), potassium (100 mEq) and calcium (800 mg). Subjects will receive supplementary high salt broth packets to ensure that they are reaching the target Na+ intake. After completion of this diet for 6 days, the subject returns to Center for Clinical Investigation - Ambulatory Clinical Center and after remaining supine for 60-90 minutes again will have blood samples obtained for future analyses and will have their blood pressure measured using an automatic recording sphygmomanometer. Readings will be obtained every 2 minutes for 20 minutes with the highest and lowest values discarded and the rest averaged. From the morning of the 6th to the morning of the 7th day, a 24-hr. urine will be collected for creatinine and sodium as a check on balance and stored for future analyses.
12. Home seated, morning cuff blood pressure and pulse will be obtained daily and monitored by study staff weekly as a safety check with the information provided to the study staff by email or phone. A member of the research team will contact the subject if the blood pressure data are not received within 24-hr of the designated time. If the cuff blood pressure is greater than 170/109 mmHg on two consecutive occasions 24 hours apart, or the subject develops cardiovascular symptoms, the subject will be terminated from the study and re-started on medications used before the washout period. The subject's physician will be contacted.
13. Because eplerenone may increase Serum K+ levels, we will monitor its level monthly during the study. This will be obtained at the time of their monthly visit unless a dose increase is made at the time of the visit. Then, the Serum K+ will be obtain one week later. If Serum K+ is greater than 5.5 mM on two consecutive occasions 24 hours apart, the subject will be terminated from the study. If unexpected adverse event is noted The Brigham and Women's Hospital Investigational Drug Pharmacy Service will be notified so as to break code and identify agent.
14. At the end of the study, twelve weeks after randomization, subjects will be counseled regarding liberal salt dietary intake. Subjects will be given high salt broth packets, calcium tablets (as calcium bicarbonate), and potassium tablets (as potassium bicarbonate) to supplement their diet to ensure similar intakes in all subjects [Na+ (200 mEq), potassium (K+, 100 mEq) and calcium (800 mg)]. This or a greater level of Na+ intake was consumed by 60-70% of subjects before entering the HyperPATH protocol. On the morning of the 6th day the subject will begin a 24-hour blood pressure recording, using a blood pressure machine provided by study staff. After completion of this diet for 6 days, the subject will come to the Center for Clinical Investigation (CCI) Ambulatory Clinical Center and after remaining supine for 60-90 mins will have blood samples obtained for future analyses, and their BP measured using an automatic recording sphygmomanometer (Space Labs, Snoqualmie, WA). Readings will be obtained every 2 mins for 20 mins with the highest and lowest values discarded and the rest averaged. From the morning of the 6th to the morning of the 7th day, a 24-hr. urine will be collected for creatinine and Na+ as a check on balance and stored for future analyses.
15. The subject then will have completed the study and will be re-started on medications used before the washout period. The subject's physician will be contacted.

ELIGIBILITY:
The subjects evaluated in this protocol are hypertensive and carry the Striatin rs254093 risk allele or both Striatin rs888083 and rs6744560 risk alleles. Most will be recruited from the HyperPATH cohort. The HyperPATH cohort was developed under a Specialized Center of Research (SCOR) in Hypertension program. This program has demographic data and DNA on more than 4000 subjects. Currently, nearly 2000 of them have undergone an extensive phenotyping protocol. All hypertensive medications have been stopped for 4 weeks before study except agents that interfere with the renin-angiotensin-aldosterone system (RAAS) are stopped for three months and amlodipine and/or hydrochlorothiazide is added if necessary for blood pressure control until one month before study initiation. Then each subject is studied twice on a diet consisting of 100 mmol potassium, 800 mg calcium, isocaloric, 2500 ml. The two times they are studied are after one week of a liberal sodium diet (200 mmol) and after one week of a low sodium diet (10 mmol). Blood is obtained supine, upright and after a 3 ng Ang II infusion and a norepinephrine dose response curve. BP and renal plasma flow are assessed in response to the diet and the Ang II infusion and 24 hour urines are collected on each diet. An oral glucose tolerance test is performed on each subject and blood is obtained for DNA. In addition to hypertensives, the nearly 2000 intensively studied cohort consists of 75 individuals in 10 families, 225 sibling pairs with hypertension, 525 normotensive individuals without a family history of hypertension or diabetes before the age of 60, and 250 type II diabetic subjects with or without hypertension. On most of the 4000 subjects serum, plasma, urine and DNA is available for measurements and analyses. Currently the data set consists of approximately 2100 data points of demographic data, family history, biomarkers, and genotypes. The subjects have been recruited from Boston, Massachusetts, Salt Lake City,ance, Rome, Italy, and Nashville Utah, Paris, Fr, Tenessee. The demographics consists of the following: 52% male, 18% of African descent, 3% Asian descent, age 17-66, hypertension stage 1-2, diet or oral medication controlled diabetes (80% of the total diabetics). A few subjects will be recruited from advertisements on the Internet and in local newspapers, from fliers and postings in the hospital, through mailings to households located in the Boston areas and through patient registries at Brigham and Womens Hospital. As an example of the richness of these sources is the Research Patient Data Registry (RPDR). RPDR is a centralized clinical data registry of 2.8 million Brigham and Womens Hospital and Massachusetts General Hospital patients. With approval of the Institutional Review Board, investigators may use the RPDR Data Acquisition Engine to obtain medical record information for patients with a specific diagnosis. Patients who meet inclusion criteria for a specific study can be identified. Potential research subjects may be contacted by his/her physician to inform the patient of the possibility of participating in a research study and to provide the patient with the information for contacting the study personnel. Investigators from Brigham and Womens Hospital may apply to use the RPDR. RPDR contains over 90,000 hypertensives, ages 17-65 years with 13.5 % of African descent and 52.8 % women.

We reported in our studies using the HyperPATH cohort that there was no racial, age or ethnic differences in the salt sensitive blood pressure responses related to Striatin allele variants. Thus, an equal number of females and males and the same proportion of Africans as in the HyperPATH cohort will be studied. Subjects in HyperPATH and those recruited for the new study in this project will have the similar characteristics. The range in age is >17; however, it is anticipated that the clear majority will be between the ages of 40 and 60 years.

Hypertensive patients previously treated will be weaned off medications for two-four weeks except agents that interfere with the renin-angiotensin-aldosterone system (RAAS) are stopped for three months and amlodipine and/or hydrochlorothiazide is added if necessary for blood pressure control until one month before study initiation. Thus, these subjects will match the characteristics of subjects recruited in HyperPATH. They must have a diastolic blood pressure between 95 and 105 mm Hg off medication in each of three screening visits. Subjects with diastolic blood pressures greater than 105 mm Hg or systolic blood pressures greater than 180 mm Hg will be excluded. Subjects with only elevated systolic blood pressure (but diastolic less than 95 mm Hg) will be excluded because such subjects were not in the HyperPATH cohort.

Based on individual statements, subjects with current excessive alcohol use (greater than 12 oz/ethanol/week) or recreational drug use will be excluded. Subjects taking other medications (except thyroid supplements) or weighing more than 150% of an ideal body weight will be excluded. Subjects with other major cardiovascular diseases, diabetes, asthma, or other major medical illness will be excluded. Subjects who smoke will be excluded. In addition, subjects must have normal values for the following screening tests: complete blood cell count (CBC), serum electrolytes, liver enzymes, Thyroid stimulating hormone (TSH), urinalysis, 24-hour urine excretion of catecholamines and cortisol, and ECG. Specifically, estimated glomerular filtration rate (GFR) must be > 60 ml/min and serum potassium < 5.0 mmol/l. Subjects with hypokalemia while on diuretics will be evaluated for hyperaldosteronism before inclusion in this study. Cushings syndrome will be ruled out clinically, and with a 24-hour urine cortisol if there is clinical uncertainty. For the more difficult question of renal artery stenosis, we will perform renal artery digital subtraction angiogram in patients with hypertension and a two-component abdominal bruit. Patients with greater than 50% renal artery stenosis will be further evaluated, but excluded from this study. Subjects with a known sensitivity to any of the agents, such as amlodipine or eplerenone will be excluded. Women who are pregnant will be excluded and will be dropped from the study if they become pregnant during the study because eplerenone has not been approved for use in pregnancy and the activity of the RAAS is dramatically altered by pregnancy.

The screened, eligible hypertensives will enter a two-week single blind placebo washout phase. Pill count will be used to determine compliance. Those with BP between 145-170/90-109 mmHg and pill count between 80-100% will enter the randomized phase, counseled regarding salt intake, and randomized double blindly into one of our two treatment arms. We will recruit approximately 105 individuals to have 45 individuals in each drug group for analyses. This assumes that we will have 10-15% non-completers.

INCLUSION CRITERIA:

1. Striatin SNP rs2540923 allele carrier OR both Striatin SNP rs888083 and Striatin SNP rs6744560 risk allele carrier
2. ages >17 years;
3. hypertension as defined by primary physician;
4. not on more than two anti-hypertensives;
5. normal renal, metabolic, electrolyte, complete blood cell count, and lipid profile laboratory tests;
6. if on an angiotensin converting enzyme inhibitor, angiotensin receptor blocker or mineralocorticoid receptor antagonist, needs to be washed out for 3 months.

EXCLUSION CRITERIA:

1. known cardiac disease other than hypertension
2. renal, circulatory or neurologic diseases
3. diabetes; smoking
4. secondary hypertension as indicated by history, physical examination or screening blood and urine tests; any drug therapy, except for anti-hypertensives and replacement thyroid medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon H Williams, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coutinho P, Vega C, Pojoga LH, Rivera A, Prado GN, Yao TM, Adler G, Torres-Grajales M, Maldonado ER, Ramos-Rivera A, Williams JS, Williams G, Romero JR. Aldosterone's rapid, nongenomic effects are mediated by striatin: a modulator of aldosterone's effect on estrogen action. Endocrinology. 2014 Jun;155(6):2233-43. doi: 10.1210/en.2013-1834. Epub 2014 Mar 21. PMID 24654783
- [Result] Garza AE, Rariy CM, Sun B, Williams J, Lasky-Su J, Baudrand R, Yao T, Moize B, Hafiz WM, Romero JR, Adler GK, Ferri C, Hopkins PN, Pojoga LH, Williams GH. Variants in striatin gene are associated with salt-sensitive blood pressure in mice and humans. Hypertension. 2015 Jan;65(1):211-217. doi: 10.1161/HYPERTENSIONAHA.114.04233. Epub 2014 Nov 3. PMID 25368024
- [Result] Pojoga LH, Coutinho P, Rivera A, Yao TM, Maldonado ER, Youte R, Adler GK, Williams J, Turchin A, Williams GH, Romero JR. Activation of the mineralocorticoid receptor increases striatin levels. Am J Hypertens. 2012 Feb;25(2):243-9. doi: 10.1038/ajh.2011.197. Epub 2011 Nov 17. PMID 22089104
- [Result] Garza AE, Pojoga LH, Moize B, Hafiz WM, Opsasnick LA, Siddiqui WT, Horenstein M, Adler GK, Williams GH, Khalil RA. Critical Role of Striatin in Blood Pressure and Vascular Responses to Dietary Sodium Intake. Hypertension. 2015 Sep;66(3):674-80. doi: 10.1161/HYPERTENSIONAHA.115.05600. Epub 2015 Jul 13. PMID 26169051
- [Result] Baudrand R, Pojoga LH, Romero JR, Williams GH. Aldosterone's mechanism of action: roles of lysine-specific demethylase 1, caveolin and striatin. Curr Opin Nephrol Hypertens. 2014 Jan;23(1):32-7. doi: 10.1097/01.mnh.0000436543.48391.e0. PMID 24275769
- [Result] Vaidya A, Underwood PC, Hopkins PN, Jeunemaitre X, Ferri C, Williams GH, Adler GK. Abnormal aldosterone physiology and cardiometabolic risk factors. Hypertension. 2013 Apr;61(4):886-93. doi: 10.1161/HYPERTENSIONAHA.111.00662. Epub 2013 Feb 11. PMID 23399714
- [Result] Brown JM, Williams JS, Luther JM, Garg R, Garza AE, Pojoga LH, Ruan DT, Williams GH, Adler GK, Vaidya A. Human interventions to characterize novel relationships between the renin-angiotensin-aldosterone system and parathyroid hormone. Hypertension. 2014 Feb;63(2):273-80. doi: 10.1161/HYPERTENSIONAHA.113.01910. Epub 2013 Nov 4. PMID 24191286
- [Result] Baudrand R, Pojoga LH, Vaidya A, Garza AE, Vohringer PA, Jeunemaitre X, Hopkins PN, Yao TM, Williams J, Adler GK, Williams GH. Statin Use and Adrenal Aldosterone Production in Hypertensive and Diabetic Subjects. Circulation. 2015 Nov 10;132(19):1825-33. doi: 10.1161/CIRCULATIONAHA.115.016759. Epub 2015 Oct 2. PMID 26432671
- [Result] Bentley-Lewis R, Adler GK, Perlstein T, Seely EW, Hopkins PN, Williams GH, Garg R. Body mass index predicts aldosterone production in normotensive adults on a high-salt diet. J Clin Endocrinol Metab. 2007 Nov;92(11):4472-5. doi: 10.1210/jc.2007-1088. Epub 2007 Aug 28. PMID 17726083
- [Result] Garg R, Williams GH, Hurwitz S, Brown NJ, Hopkins PN, Adler GK. Low-salt diet increases insulin resistance in healthy subjects. Metabolism. 2011 Jul;60(7):965-8. doi: 10.1016/j.metabol.2010.09.005. Epub 2010 Oct 30. PMID 21036373
- [Result] Pojoga LH, Underwood PC, Goodarzi MO, Williams JS, Adler GK, Jeunemaitre X, Hopkins PN, Raby BA, Lasky-Su J, Sun B, Cui J, Guo X, Taylor KD, Chen YD, Xiang A, Raffel LJ, Buchanan TA, Rotter JI, Williams GH. Variants of the caveolin-1 gene: a translational investigation linking insulin resistance and hypertension. J Clin Endocrinol Metab. 2011 Aug;96(8):E1288-92. doi: 10.1210/jc.2010-2738. Epub 2011 May 25. PMID 21613355
- [Result] Underwood PC, Sun B, Williams JS, Pojoga LH, Chamarthi B, Lasky-Su J, Raby BA, Hopkins PN, Jeunemaitre X, Brown NJ, Adler GK, Williams GH. The relationship between peroxisome proliferator-activated receptor-gamma and renin: a human genetics study. J Clin Endocrinol Metab. 2010 Sep;95(9):E75-9. doi: 10.1210/jc.2010-0270. Epub 2010 Jul 14. PMID 20631015
- [Result] Underwood PC, Sun B, Williams JS, Pojoga LH, Raby B, Lasky-Su J, Hunt S, Hopkins PN, Jeunemaitre X, Adler GK, Williams GH. The association of the angiotensinogen gene with insulin sensitivity in humans: a tagging single nucleotide polymorphism and haplotype approach. Metabolism. 2011 Aug;60(8):1150-7. doi: 10.1016/j.metabol.2010.12.009. Epub 2011 Feb 8. PMID 21306748
- [Result] Pojoga LH, Romero JR, Yao TM, Loutraris P, Ricchiuti V, Coutinho P, Guo C, Lapointe N, Stone JR, Adler GK, Williams GH. Caveolin-1 ablation reduces the adverse cardiovascular effects of N-omega-nitro-L-arginine methyl ester and angiotensin II. Endocrinology. 2010 Mar;151(3):1236-46. doi: 10.1210/en.2009-0514. Epub 2010 Jan 22. PMID 20097717
- [Result] Chong C, Hamid A, Yao T, Garza AE, Pojoga LH, Adler GK, Romero JR, Williams GH. Regulation of aldosterone secretion by mineralocorticoid receptor-mediated signaling. J Endocrinol. 2017 Mar;232(3):525-534. doi: 10.1530/JOE-16-0452. Epub 2017 Jan 17. PMID 28096435
- [Result] Pojoga LH, Yao TM, Sinha S, Ross RL, Lin JC, Raffetto JD, Adler GK, Williams GH, Khalil RA. Effect of dietary sodium on vasoconstriction and eNOS-mediated vascular relaxation in caveolin-1-deficient mice. Am J Physiol Heart Circ Physiol. 2008 Mar;294(3):H1258-65. doi: 10.1152/ajpheart.01014.2007. Epub 2008 Jan 4. PMID 18178722
- [Derived] Stone IB, Green JAEM, Koefoed AW, Hornik ES, Williams JS, Adler GK, Williams GH. Striatin genotype-based, mineralocorticoid receptor antagonist-driven clinical trial: study rationale and design. Pharmacogenet Genomics. 2021 Jun 1;31(4):83-88. doi: 10.1097/FPC.0000000000000425. PMID 33904521

RESULTS

PARTICIPANT FLOW:
Groups:
- Epleronone Arm: The first dose was 50mg/day; the second dose was 100mg /day, and the third dose was 200 mg/day. Eplerenone vs Amlodipine: We posit that decreases in striatin activity/levels increases aldosterone secretion resulting in hypertension and salt sensitive blood pressure. Thus, our mechanistic clinical study will assess whether hypertensive striatin risk allele carriers will show significantly greater reductions in blood pressure with a specific aldosterone mediated treatment approach (mineralocorticoid receptor blockade) than with a non-specific approach (amlodipine). To test this hypothesis, we will perform a randomized, double-blind, active controlled study in hypertensive carriers of the striatin risk allele using a novel two-limb, proof-of-principle study. Our primary outcome will be a liberal salt diet systolic blood pressure with a secondary outcome of salt sensitive blood pressure. Therefore, this mechanistic trial will provide support for using a genetic marker that identifies individuals who are uniquely responsive to mineralocorticoid receptor blockade--personalized, precision medicine.
- Amlodipine Arm: Starting Dose for Amlodipine 2.5 mg/day; Second Dose is 5.0 mg/day; the Third Dose was 10 mg/day. Eplerenone vs Amlodipine: We posit that decreases in striatin activity/levels increases aldosterone secretion resulting in hypertension and salt sensitive blood pressure. Thus, our mechanistic clinical study will assess whether hypertensive striatin risk allele carriers will show significantly greater reductions in blood pressure with a specific aldosterone mediated treatment approach (mineralocorticoid receptor blockade) than with a non-specific approach (amlodipine). To test this hypothesis, we will perform a randomized, double-blind, active controlled study in hypertensive carriers of the striatin risk allele using a novel two-limb, proof-of-principle study. Our primary outcome will be a liberal salt diet systolic blood pressure with a secondary outcome of salt sensitive blood pressure. Therefore, this mechanistic trial will provide support for using a genetic marker that identifies individuals who are uniquely responsive to mineralocorticoid receptor blockade--personalized, precision medicine.
Period: Overall Study
Arm/Group | Epleronone Arm | Amlodipine Arm
Started | 45 | 45
Completed | 33 (Coronavirus Disease 2019 (COVID-19) delayed and funds ended) | 32 (Coronavirus Disease 2019 (COVID-19) delayed and funds ended)
Not Completed | 12 | 13
Not completed — see limitations | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Epleronone Arm; Amlodipine Arm: Eplerenone vs Amlodipine: We posit that decreases in striatin activity/levels increases aldosterone secretion resulting in hypertension and salt sensitive blood pressure. Thus, our mechanistic clinical study will assess whether hypertensive striatin risk allele carriers will show significantly greater reductions in blood pressure with a specific aldosterone mediated treatment approach (mineralocorticoid receptor blockade) than with a non-specific approach (amlodipine). To test this hypothesis, we will perform a randomized, double-blind, active controlled study in hypertensive carriers of the striatin risk allele using a novel two-limb, proof-of-principle study. Our primary outcome will be a liberal salt diet systolic blood pressure with a secondary outcome of salt sensitive blood pressure. Therefore, this mechanistic trial will provide support for using a genetic marker that identifies individuals who are uniquely responsive to mineralocorticoid receptor blockade--personalized, precision medicine.
- Total: Total of all reporting groups
Arm/Group | Epleronone Arm | Amlodipine Arm | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 32 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (8.6) | 53.8 (10.1) | 55 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 29 | 31 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 12 | 22
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65
body mass index [Mean (Standard Deviation); unit: kg/m squared] | 30.0 (6.2) | 31.5 (3.8) | 30.7 (6.3)
systolic blood pressure [Mean (Standard Deviation); unit: mm hg] | 144.2 (15) | 148.5 (10.5) | 146.4 (15.3)
diastolic blood pressure [Mean (Standard Deviation); unit: mm hg] | 86.0 (7.7) | 91.4 (7.2) | 88.5 (7.8)
Salt Sensitivity of Blood Pressure (SSBP) systolic [Mean (Standard Deviation); unit: mm hg] | 8.6 (13.6) | 11.1 (10.9) | 9.9 (13.7)
SSBP diastolic [Mean (Standard Deviation); unit: mm hg] | 3.5 (7.6) | 4.5 (7.5) | 4.0 (7.7)
HGBA1C [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 5.4 (0.4) | 5.4 (0.3) | 5.4 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Systolic /Diastolic Supine Morning Liberal Salt Automated Blood Pressure
Description: Subjects will be counseled regarding liberal salt dietary intake to ensure similar intakes in all subjects [Na+ (200 mEq), potassium (K+, 100 mEq) and calcium (800 mg)]. This or a greater level of Na+ intake was consumed by 60-70% of subjects before entering the International Hypertensive Pathotype (HyperPATH) protocol. After completion of this diet for 7 days, the subject will come to the Center for Clinical Investigation (CCI) Ambulatory Clinical Center between 7-8 morning (AM), fasting, and after remaining supine for 60-90 mins will have blood samples obtained for future analyses, and their BP measured using an automatic recording sphygmomanometer. Readings will be obtained every 2 mins for 20 mins with the highest and lowest values discarded and the rest averaged. From the morning of the 6th to the morning of the 7th day, a 24hr. urine will be collected for creatinine and Na+ as a check on balance and stored for future analyses. Procedure will be performed before randomization and
Time Frame: Change in blood pressure between visit 2 (baseline), visit 3 (four weeks), visit 4 (8 weeks), visit 5 (12 weeks) of randomized drug therapy
Population: baseline liberal salt diet
Measure: Mean (Standard Deviation); unit: mm hg
Arm/Group | Epleronone Arm | Amlodipine Arm
Number analyzed (Participants) | 33 | 32
mm hg
  visit 2 systolic bp | 144.2 (15) | 148.5 (10.5)
  visit 2 diastolic bp | 86.0 (7.7) | 91.4 (7.2)
  visit 3 systolic bp | 137.1 (13.2) | 144.5 (12.1)
  visit 3 diastolic bp | 83.7 (8.1) | 90.8 (7.8)
  visit 4 systolic bp | 135.4 (13.9) | 140.7 (11.8)
  visit 4 diastolic bp | 82.8 (8.4) | 87.5 (7.5)
  visit 5 Systolic BP | 134.3 (11.7) | 135.9 (12.1)
  Visit 5 diastolic bp | 83.1 (7.6) | 85.9 (7.7)
Statistical Analysis 1: Comparison: Epleronone Arm vs Amlodipine Arm; adjusted to medication dose, sex, age, race; Test type: Superiority; p = 0.823, Regression, Linear
Statistical Analysis 2: Comparison: Epleronone Arm; diastolic bp adjusted for medication dose sex,age, race; Test type: Superiority; p = .8390, Regression, Linear

2. Primary Outcome: Systolic/Diastolic Blood Pressure Visit 2, 3, 4, 5 Eplerenone vs Amlodipine
Description: First step: subjects will ingest a liberal salt intake [Na+ (200 mEq/day)] for 7 days. The subject will come to the study unit between 7-8 AM, fasting. After remaining supine for 60-90 mins, their BP will be measured using an automatic recording sphygmomanometer. Readings will be obtained every 2 mins for 20 mins with the highest and lowest values discarded and the rest averaged. From the morning of the 6th to the morning of the 7th day, a 24-hr. urine will be collected for creatinine and Na+ as a check on balance and stored for future analyses. Second step: subjects will then be fed a restricted salt diet (10 mEq Na+/day) for 7 days. On the morning of the 7th day, the subjects will come fasting to the study unit between 7-8 AM, and the studies performed as detailed above. The BP data from the two diet studies will allow us to calculate SSBP. The procedures will be performed before randomization and at the completion of 12 weeks of therapy.
Time Frame: Change in blood pressure between eplerenone and amlodipine at visit 2 (baseline), visit 3 (four weeks), visit 4 (8 weeks), visit 5 (12 weeks) of randomized drug therapy
Measure: Mean (Standard Deviation); unit: mm hg
Arm/Group | Epleronone Arm | Amlodipine Arm
Number analyzed (Participants) | 33 | 32
mm hg
  visit 2 systolic | 144.2 (15) | 148.5 (10.5)
  visit2 diastolic | 86.0 (7.7) | 91.4 (7.2)
  systolic visit 3 | 137.1 (13.2) | 144.5 (12.1)
  visit 3 diastolic | 83.7 (8.1) | 90.8 (7.8)
  visit 4 systolic | 135.4 (13.9) | 140.7 (11.8)
  visit 4 diastolic | 82.8 (8.4) | 87.5 (7.5)
  visit 5 systolic | 134.3 (11.7) | 135.9 (12.1)
  visit 5 diastolic | 83.1 (7.6) | 85.9 (7.7)
Statistical Analysis 1: Comparison: Epleronone Arm vs Amlodipine Arm; Test type: Superiority; p = .0101, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: 24 hr bp
Description: For this measurement, we used a separate set of data - continuous monitoring of blood pressure. These blood pressure measurements are different than those reported in the Primary Outcomes section. The Secondary Outcomes are continuous 24-hour blood pressures, measured twice. The 24 hour assessment was divided into 3 sections: total 24-hour, daytime and night; Change in blood pressure between visit 2 (baseline) and visit 5 (12 weeks) of randomized drug therapy
Time Frame: total 24 hour, daytime and night Change in blood pressure between visit 2 (baseline) and visit 5 (12 weeks) of randomized drug therapy
Measure: Mean (Standard Deviation); unit: mm hg
Arm/Group | Epleronone Arm | Amlodipine Arm
Number analyzed (Participants) | 33 | 31
mm hg
  24 hr systolic | 8.45 (11.89) | 9.9 (10.28)
  24 hour diastolic | 4.33 (7.88) | 5.41 (6.73)
  awake systolic | 7.69 (13.15) | 10.03 (12.31)
  awake diastolic | 4.09 (9.02) | 5.35 (7.67)
  asleep systolic | 8.72 (13.01) | 10.96 (9.94)
  asleep diastolic | 3.63 (10.12) | 6.16 (7.4)
Statistical Analysis 1: Comparison: Epleronone Arm vs Amlodipine Arm; Test type: Superiority; p = 0.59, ANOVA

4. Other Pre Specified Outcome: The Percent of Individuals Who Achieved Goal Blood Pressure (e.g., <140/90 mmHg) at Each Time
Description: We analyzed our results using Kaplan-Meier Plot and Cox-Hazard ratios and used the number of subjects who achieved goal blood pressure (e.g., <140/90 mmHg) at weeks 0 (visit 2), 4 (Visit 3), 8 Visit 4), 12 (Visit 5), and Number that did not achieve goal BP at Visit 5 (week 12). Those individuals at week 12 who did not achieve goal blood pressure were identified as a separate group and termed non-responders. Thus, the value at each time is the percent of subjects at that time who achieved goal blood pressure.
Time Frame: Those who achieved goal blood pressure at weeks 0 (visit 2), 4 (Visit 3), 8 Visit 4), 12 (Visit 5), and Number that did not achieve goal BP at Visit 5 (week 12). of randomized drug therapy
Population: all subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Epleronone Arm | Amlodipine Arm
Number analyzed (Participants) | 33 | 32
Participants
  Visit 2 (week 0) | 33 | 32
  Visit 3 (week 4) | 13 | 7
  Visit 4 (week 8) | 6 | 4
  Visit 5 (week 12) | 7 | 10
  Number that did not achieve goal BP at Visit 5 (week 12) | 7 | 11
Statistical Analysis 1: Comparison: Epleronone Arm vs Amlodipine Arm; Test type: Superiority; p = .09, Kaplan-Meier using Gehan-Breslow-Wilcoxo; Hazard Ratio, log = .7022

ADVERSE EVENTS:
Time Frame: 120 days
Arm/Group | Epleronone Arm | Amlodipine Arm
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 3/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epleronone Arm (N=33) | Amlodipine Arm (N=32)
swelling (General disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Early termination of the trial was secondary to the adverse effects of the Coronavirus Disease 2019 (COVID-19) pandemic. 1. We were shut down for 8 months in 2020-21. 2. Enrolled, not completed subjects, had to begin the study again. 3. Recruiting new subjects during the pandemic was extremely difficult. 4. NIH funded the trial, but no additional funds were available to cover the short fall. Further studies will be required to determine if the hypothesis being tested is correct.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT03683069/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT03683069/SAP_001.pdf